CLINICAL TRIAL: NCT01374542
Title: Respiratory Endoscopy: Diagnostic Yield, Technical Factors and Complications
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/350/C
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Lung Neoplasm; Lung Diseases, Interstitial; Respiratory Tract Infections; Pleural Effusions
Keywords: Bronchoscopy; Thoracoscopy
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases, Interstitial; Respiratory Tract Infections; Pleural Effusion | interventions — Thoracoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Respiratory endoscopy patients: Patients undergoing respiratory endoscopy at Singapore General Hospital
  Interventions: Procedure: Respiratory endoscopy

INTERVENTIONS:
Procedure: Respiratory endoscopy — Bronchoscopy, thoracoscopy, endobronchial ultrasound
  Other Names: Bronchoscopy-Flexible bronchoscopy; Thoracoscopy-Pleuroscopy; Endobronchial ultrasound-EBUS

SUMMARY:
Background: Respiratory endoscopy comprises flexible bronchoscopy and medical thoracoscopy. The diagnostic yield, technical factors and complications for all patient sub-populations is still not clearly defined. This may result in inappropriate or even dangerous application of such procedures. The aim of the study is to collect data on these aspects of respiratory endoscopy and identify important trends, as well as, areas for improvement. This data will also provide baseline comparative data for new bronchoscopic techniques such as endobronchial ultrasound and navigational bronchoscopy.

Method: Prospective data collection. Technical details regarding these procedures are currently keyed into the OTM system by the endoscopy operators for documentation and billing. The department of Respiratory and Critical Care Medicine gets monthly downloads of all the fields from the OTM system for audit purposes.(See data collection form) The research project proposes to make the data non identifiable by removing the patient's name and IC number. Additionally the yield of the procedure will be checked by a chart review of the histology and microbiology results. There are no restrictions on patient recruitment because all procedures will be performed for clinical indications only and no patient will be recruited for the sole purpose of the study. Waiver of consent has been approved by the IRB.

DETAILED DESCRIPTION:
Background: Respiratory endoscopy comprises flexible bronchoscopy and medical thoracoscopy. The diagnostic yield, technical factors and complications for all patient sub-populations is still not clearly defined. This may result in inappropriate or even dangerous application of such procedures. The aim of the study is to collect data on these aspects of respiratory endoscopy and identify important trends, as well as, areas for improvement. This data will also provide baseline comparative data for new bronchoscopic techniques such as endobronchial ultrasound and navigational bronchoscopy.

Method: Prospective data collection. Technical details regarding these procedures are currently keyed into the OTM system by the endoscopy operators for documentation and billing. The department of Respiratory and Critical Care Medicine gets monthly downloads of all the fields from the OTM system for audit purposes.(See data collection form) The research project proposes to make the data non identifiable by removing the patient's name and IC number. Additionally the yield of the procedure will be checked by a chart review of the histology and microbiology results. There are no restrictions on patient recruitment because all procedures will be performed for clinical indications only and no patient will be recruited for the sole purpose of the study. Waiver of consent has been obtained by the IRB. The current estimated bronchoscopy load is 1000/year and data will be kept in the trial co-coordinator's computer in a locked office. The investigators hope to run the database for 3 years initially.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing respiratory endoscopy at Singapore General Hospital

Exclusion Criteria:

* Clinical contra-indications to respiratory endoscopy

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing respiratory endoscopy at Singapore General Hospital
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2011-06; Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Endoscopy diagnostic yield | 1 year
  Positive and negative histology and microbiology yield
Endoscopy technical factors | 1 year
  Duration, sedation requirements, consumables
Endoscopy safety | 1 year
  Complication rate, need for escalation of care

CONTACTS AND LOCATIONS:
Overall Officials: Devanand Anantham, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Kawaraya M, Gemba K, Ueoka H, Nishii K, Kiura K, Kodani T, Tabata M, Shibayama T, Kitajima T, Tanimoto M. Evaluation of various cytological examinations by bronchoscopy in the diagnosis of peripheral lung cancer. Br J Cancer. 2003 Nov 17;89(10):1885-8. doi: 10.1038/sj.bjc.6601368. PMID 14612897
- [Background] Torrington KG, Kern JD. The utility of fiberoptic bronchoscopy in the evaluation of the solitary pulmonary nodule. Chest. 1993 Oct;104(4):1021-4. doi: 10.1378/chest.104.4.1021. PMID 8404158
- [Derived] Quek JC, Tan QL, Allen JC, Anantham D. Malignant pleural effusion survival prognostication in an Asian population. Respirology. 2020 Dec;25(12):1283-1291. doi: 10.1111/resp.13837. Epub 2020 May 11. PMID 32390227
- [Derived] Choo R, Naser NSH, Nadkarni NV, Anantham D. Utility of bronchoalveolar lavage in the management of immunocompromised patients presenting with lung infiltrates. BMC Pulm Med. 2019 Feb 26;19(1):51. doi: 10.1186/s12890-019-0801-2. PMID 30808314
- [Derived] De Roza MA, Quah KH, Tay CK, Toh W, Li H, Kalyanasundaram G, Anantham D. Diagnosis of Peripheral Lung Lesions via Conventional Flexible Bronchoscopy with Multiplanar CT Planning. Pulm Med. 2016;2016:5048961. doi: 10.1155/2016/5048961. Epub 2016 Nov 13. PMID 27957340